CLINICAL TRIAL: NCT03766737
Title: Validation of the Utility of an Intelligent Visual Acuity Diagnostic System for Children: Using a Human-in-the-loop Artificial Intelligence Paradigm
Brief Title: Validation of the Utility of an Intelligent Visual Acuity Diagnostic System for Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CCPMOH2018-China-12
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Ophthalmopathy; Artificial Intelligence
Keywords: Vision Disorders
MeSH Terms: conditions — Eye Diseases; Vision Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eligible patients for AI test. (Other): Device: An intelligent visual acuity diagnostic system for children. An artificial intelligence to evaluate children's vision.
  Interventions: Device: An intelligent visual acuity diagnostic system for children

INTERVENTIONS:
Device: An intelligent visual acuity diagnostic system for children — An artificial intelligence to make evaluation and of children's vision.

SUMMARY:
Visual development during early childhood is a vital process. Examining the visual acuity of children is essential for the early detection of visual abnormality, but performing such an assessment in children is challenging. Here, the investigators developed a human-in-the-loop artificial intelligence (AI) paradigm that combines traditional vision examination and AI with integrated software and hardware, thus making the vision examination easy to perform. The investigator also establish a entity intelligent visual acuity diagnostic system based on the paradigm, and conduct clinical trial to validate if the diagnostic system can offsetting the shortcomings of human doctors.

ELIGIBILITY:
Inclusion Criteria:

* Paediatric patients from eye clinic written informed consents provided

Ages: 1 Month to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2018-05-20 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
The proportion of accurate, mistaken and miss detection of the intelligent visual acuity diagnostic system. | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lin Haotian, M.D, Ph.D, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China